CLINICAL TRIAL: NCT04955899
Title: A Single Arm Pilot Study to Evaluate the Safety and Feasibility of Splenic Nerve Stimulation in Patients With Rheumatoid Arthritis Using an Active Implantable Device
Brief Title: Safety of Splenic Stimulation for RA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galvani Bioelectronics (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GAL1039
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Electrical stimulation; inflammation; active implantable medical device; Laparoscopy; antirheumatic agents; autonomic nervous system; feasibility studies
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Stimulation (Experimental): Active stimulation for 12 weeks
  Interventions: Device: Active Stimulation

INTERVENTIONS:
Device: Active Stimulation — The Galvani System will be implanted in eligible participants, and stimulation will be turned ON

SUMMARY:
This study will evaluate the safety and tolerability of stimulating the splenic neurovascular bundle (NVB) with the Galvani System, which consists of a lead, implantable pulse generator, external components and accessories. Participants eligible for implant will have active rheumatoid arthritis (RA) and have an inadequate response or intolerance to at least two biologic Disease Modifying Anti-Rheumatic Drugs (DMARDs) or JAK inhibitors (JAKis). Five participants will be implanted with the device and receive neurostimulation for 12 weeks.

DETAILED DESCRIPTION:
The study will be an open-label single-arm study to evaluate the safety and tolerability of Galvani's neuromodulation system. Participants with active rheumatoid arthritis (RA) will be implanted with the Galvani system and receive active stimulation for 12 weeks. The total study duration in the study for each participant is approximately 5 months, with a 4-week screening period, 4 weeks recovery from surgery and a 12-week 'treatment' period. The participants will return to the clinic on pre-defined days for follow-up visits during the trial period. At Days 42 and/or Day 56, if study participants are not responding to stimulation, stimulation parameters might be adapted. At the end of the study (Day-84), participants will enroll in a long-term follow-up study up to 5-years after enrollment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset RA of at least six months duration
* Male or female participants, 22-75 years of age
* Active RA
* Inadequate Response to at least 2 biologic DMARDs and/or JAK- inhibitors (JAKis)
* Have an appropriate washout from previously used biological DMARDs or JAKi
* A female participant should have no child-bearing potential

Exclusion Criteria:

* Inability to provide informed consent.
* Significant psychiatric disease or substance abuse.
* History of unilateral or bilateral vagotomy.
* Active or latent tuberculosis
* Known infection with human immunodeficiency virus (HIV); current acute or chronic hepatitis B or hepatitis C; previous hepatitis B.
* Currently implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators).
* Previous splenectomy
* Any investigational small molecule drug or biological within 2 weeks or 2 half-lives whichever is longer, before surgery.
* Uncontrolled other inflammatory diseases
* Current/recurrent infections that in the opinion of the PI risk>benefit.
* History of cancer within the past 5 years, except non-malignant skin cancer.
* Chronic use of morphine or oxicodone

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the Galvani system | 12 weeks
  Incidence and relatedness of Adverse Events (AEs), which include clinically significant findings from Laboratory Safety Assessments (clinical chemistry and hematology), vital signs (blood pressure, heart rate, respiratory rate, and body temperature), and 12-Lead ECG

SECONDARY OUTCOMES:
Effect of stimulation on the change in pharmacodynamic and response biomarkers | Day 1 to week 12
  Changes from baseline (Day 1) in the levels of LPS-inducible cytokine/ chemokine release, in whole blood assay at different timepoints after start of stimulation
To evaluate the usability of the external Galvani System devices and accessories | 12 weeks
  Summarize feedback collected on questionnaires pertaining to the use of the external Galvani System devices
To evaluate the participants' perception of therapy and sensation | 12 weeks
  Summarize feedback collected on questionnaires
Evaluate device performance | 12 weeks
  Tabulation of device deficiencies

CONTACTS AND LOCATIONS:
Locations (2):
- Academic Medical Center (AMC) Dept of Rheumatology & Clinical Immunology, Amsterdam, Netherlands
- Greater Glasgow Health Board, Glasgow, United Kingdom